CLINICAL TRIAL: NCT02654769
Title: Multicenter Randomized Double-Blind Vehicle-Controlled Parallel Group Study to Determine the Therapeutic Equivalence of Generic Ingenol Mebutate Gel 0.05% and Picato® Gel 0.05% in Subjects With Actinic Keratosis on the Trunk or Extremities
Brief Title: A Study of Equivalence of Generic Ingenol Mebutate Gel 0.05% and Picato Gel 0.05% in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 094-8151-301
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Comparator Picato® (Active Comparator): Picato® (ingenol mebutate) gel, 0.05% (Leo Pharma Inc.) [Reference Listed Drug (RLD)]
  Interventions: Drug: Ingenol Mebutate (Picato®)
- Generic Ingenol Mebutate (Experimental): Generic ingenol mebutate gel, 0.05% [Test]
  Interventions: Drug: Generic Ingenol Mebutate
- Vehicle Foam (Placebo Comparator): Vehicle gel of the test product
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Ingenol Mebutate (Picato®) — Brand product
  Other Names: Picato
  Arms: Active Comparator Picato®
Drug: Generic Ingenol Mebutate — Generic formulated to have the same therapeutic effect of the brand
  Arms: Generic Ingenol Mebutate
Drug: Vehicle Foam — It does not contain active ingredient. A placebo to test the sensitivity of the active treatments.
  Other Names: Placebo
  Arms: Vehicle Foam

SUMMARY:
The objective of this study was to evaluate the safety and therapeutic equivalence of generic ingenol mebutate gel, 0.05% to Picato gel, 0.05% and to establish the superiority of the efficacy of these two products over the vehicle gel in the treatment of Actinic Keratosis (AK) on the trunk or extremities.

DETAILED DESCRIPTION:
Picato® (ingenol mebutate) gel is the first and only ingenol mebutate product approved by the FDA in 2012 for the topical treatment of AK(s) on the face and scalp (0.015% formulation) and on the trunk and extremities (0.05% formulation). A generic ingenol mebutate gel, 0.05% has been developed for the topical treatment of clinically typical, visible, and discrete non-hyperkeratotic, non-hypertrophic AK lesions of the trunk or extremities.

ELIGIBILITY:
Inclusion Criteria:

* Subject was a male or non-pregnant female 18 years of age or older
* Subject provided written informed consent.
* Subject was willing and able to apply the test article as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
* Subject had a clinical diagnosis of AK at Baseline with at least four (4), but no more than eight (8), visible and discrete non-hyperkeratotic, non-hypertrophic AK lesions, each at least 4 mm in diameter, within a contiguous 25 cm2 treatment area ("the Treatment Area") on the trunk or extremities.
* Subject was in good general health and free of any disease state or physical condition that might have impaired evaluation of AK lesions or which, in the investigator's opinion, exposed the subject to an unacceptable risk by study participation.
* Females must have been post-menopausal , surgically sterile , or have used an effective method of birth control , with a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

* Subject was pregnant, lactating, or was planning to become pregnant during the study.
* Subject was currently enrolled in an investigational drug or device study.
* Subject used an investigational drug or investigational device treatment within 30 days prior to the Baseline Visit.
* Subject had hyperkeratotic, hypertrophic, or large mat-like AKs (e.g., AK >1 cm2 in size) within the contiguous 25 cm2 Treatment Area.
* Subject had more than eight (8) AKs, independent of size, within the contiguous 25 cm2 Treatment Area.
* Subject had the need or planned to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Subject was immunosuppressed (e.g., HIV, systemic malignancy, graft host disease, etc.)
* Subject had experienced an unsuccessful outcome from previous ingenol mebutate therapy (an unsuccessful outcome was defined as after a reasonable therapeutic trial with no compliance issues and the topical drug did not work).
* Subject had a history of sensitivity to any of the ingredients in the test articles (see Section 9.4.2).
* Subject used topical creams, lotions, or gels of any kind within the selected Treatment Area within one (1) day prior to entry into the study.
* Subject used topical medications; corticosteroids, alpha hydroxy acids (e.g., glycolic acid, lactic acid etc. >5%), beta hydroxy acid (salicylic acid >2%), urea >5%, 5-fluorouracil, diclofenac, imiquimod, ingenol mebutate, or prescription retinoids (e.g., tazarotene, adapalene, tretinoin) within the selected Treatment Area (trunk or extremities) within one (1) month prior to the Baseline Visit.
* Subject had cryodestruction, curettage, photodynamic therapy, surgical excision, or other treatments for AK within the selected Treatment Area (trunk or extremities) within one (1) month prior to the Baseline Visit.
* Subject used oral corticosteroid therapy, interferon, cytotoxic drugs, immunomodulators, immunosuppressive therapies, or retinoids within one (1) month prior to the Baseline Visit.
* Subject had dermatologic procedures or surgeries such as laser resurfacing, Psoralen + ultraviolet A (PUVA) therapy, ultraviolet B (UVB) therapy, chemical peels, or dermabrasion on the selected Treatment area (trunk or extremities) within six (6) months prior to the Baseline Visit.
* Subject had lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the selected Treatment Area (trunk or extremities).
* Subject had any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the test article or required the use of interfering topical, systemic, or surgical therapy.
* Subject had any condition which, in the investigator's opinion, would have made it unsafe or precluded the subject's ability to fully participate in this research study.
* Subject was unable to communicate or cooperate with the investigator due to language problems, poor mental development, impaired cerebral function, or physical limitations.
* Subject was known to be noncompliant or was unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.
* Subject had been previously enrolled in the same study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Khatsenko, Ph.D, Study Director — Actavis Inc.
Locations (22):
- United States (22):
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - SD Sports Medicine & Family Health Center, San Diego, California
  - The Center for Clinical and Cosmetic Research, Aventura, Florida
  - Savin Medical Group Research Center, Miami Lakes, Florida
  - Tory P. Sullivan, M.D., P.A., North Miami Beach, Florida
  - Moore Clinical Research, Inc., Tampa, Florida
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Christie Clinic, LLC, Champaign, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Bettencourt Skin Center, Henderson, Nevada
  - Union Square Dermatology, New York, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Omega Medical Research, 400 Bald Hill Road, Warwick, RI 02886, Warwick, Rhode Island
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - DermResearch, Inc.Austin, Austin, Texas
  - The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator Picato® | Generic Ingenol Mebutate | Vehicle Foam
Started | 149 | 149 | 143
Completed | 145 | 148 | 142
Not Completed | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects in Modified Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator Picato® | Generic Ingenol Mebutate | Vehicle Foam | Total
Number analyzed (Participants) | 148 | 149 | 142 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.49) | 66.6 (11.11) | 66.2 (9.07) | 66.7 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 76 | 66 | 200
  Male | 90 | 73 | 76 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 13 | 40
  Not Hispanic or Latino | 133 | 137 | 129 | 399
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 148 | 149 | 141 | 438
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Fitzpatrick Skin Type I [Count of Participants; unit: Participants] — Typical features: Pale white skin, blue/hazel eyes, blond/red hair. Tanning ability: Always burns, does not tan.
  Participants | 26 | 32 | 22 | 80
Fitzpatrick Skin Type II [Count of Participants; unit: Participants] — Typical features: fair skin, blue eyes. Tanning ability: burns easily, tans poorly.
  Participants | 63 | 56 | 67 | 186
Fitzpatrick Skin Type III [Count of Participants; unit: Participants] — Typical features: darker white skin. Tanning ability: tans after initial burn.
  Participants | 49 | 52 | 43 | 144
Fitzpatrick Skin Type IV [Count of Participants; unit: Participants] — Typical features: light brown skin. Tanning ability: burns minimally, tans easily.
  Participants | 9 | 8 | 10 | 27
Fitzpatrick Skin Type V [Count of Participants; unit: Participants] — Typical features: brown skin. Tanning ability: rarely burns, tans darkly easily.
  Participants | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Outcome Measure
Description: Percentage of subjects in the PP population in each treatment group with complete clearance of AK lesions. Complete clearance was defined as having no (zero) clinically visible AK lesions in the Treatment Area at the Week 8 visit.
Time Frame: 8 weeks
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator Picato® | Generic Ingenol Mebutate | Vehicle Foam
Number analyzed (Participants) | 131 | 135 | 132
Participants | 50 | 49 | 8
Statistical Analysis 1: Comparison: Active Comparator Picato® vs Generic Ingenol Mebutate; Test type: Equivalence — Difference (Generic- Picato); p < 0.0001, Fisher Exact; 90% Wald's confidence interval = -1.87, 90% CI 2-sided [-12.37 to 8.63]

2. Secondary Outcome: The Percentage of Subjects in the PP Population in Each Treatment Group With Partial Clearance (as Having at Least 75% Reduction in the Number of Clinically Visible AK Lesions) in theTreatment Area at the Week 8 Visit.
Time Frame: 8 weeks
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator Picato® | Generic Ingenol Mebutate | Vehicle Foam
Number analyzed (Participants) | 131 | 135 | 132
Participants | 84 | 83 | 21
Statistical Analysis 1: Comparison: Active Comparator Picato® vs Generic Ingenol Mebutate; Partial Clearance at Week 8; Test type: Equivalence — Difference (Generic - Picato); p < 0.0001, Fisher Exact; 90% Wald's confidence interval = -2.64, 90% CI 2-sided [-13.14 to 7.86]

ADVERSE EVENTS:
Time Frame: From the start of the study until Week 8 (end of study).
Arm/Group | Generic Ingenol Mebutate | Active Comparator Picato® | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/149 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/149 | 0/143
Other Adverse Events (participants affected / at risk) | 18/149 | 29/149 | 17/143
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Ingenol Mebutate (N=149) | Active Comparator Picato® (N=149) | Vehicle Foam (N=143)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Conjunctival irritation (Eye disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Application site erosion (General disorders) | 2 | 2 | 0
Application site hypoaesthesia (General disorders) | 1 | 0 | 0
Application site pain (General disorders) | 0 | 7 | 0
Application site pruritus (General disorders) | 1 | 3 | 0
Application site scab (General disorders) | 0 | 1 | 0
Application site vesicles (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Application site abscess (Infections and infestations) | 0 | 1 | 0
Application site cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Genital herpes simplex (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphyloccocall skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Hyperlipidaemis (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Spider vein (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.